CLINICAL TRIAL: NCT03303339
Title: A Phase 1b/2 Study of PCM-075 (Onvansertib) in Combination With Either Low-Dose Cytarabine or Decitabine in Subjects With Acute Myeloid Leukemia (AML)
Brief Title: Onvansertib in Combination With Either Low-dose Cytarabine or Decitabine in Adult Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROV-052; U1111-1201-6416 (Other: WHO)
Record Dates: First submitted 2017-09-06; First posted 2017-10-06 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: PLK1; PLK Inhibitor; Onvansertib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — onvansertib; Cytarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b: Onvansertib + low-dose cytarabine (Experimental): Onvansertib, administered in escalating doses orally Day 1 through Day 5 every 28 days (1 cycle) in combination with cytarabine, which will be administered in all cohorts as 20 mg/m^2 subcutaneously, once daily on Day 1 through Day 10 every 28 days (1 cycle). Onvansertib administration, in combination with cytarabine, will be initiated at a starting dose of 12 mg/m^2 orally, daily for 5 days. Onvansertib dose will be escalated in successive cohorts until the recommended phase 2 dose is achieved.
  Interventions: Drug: Onvansertib; Drug: Cytarabine
- Phase 1b: Onvansertib + decitabine (Experimental): Onvansertib will be administered in escalating doses orally, Day 1 through Day 5 every 28 days (1 cycle) in combination with decitabine, administered consistently in all cohorts as 20 mg/m^2 intravenously over 1 hour on Day 1 through Day 5 every 28 days (1 cycle). Onvansertib administration, in combination with decitabine, will be initiated at a starting dose of 12 mg/m^2 orally, daily for 5 days (Day 1 through Day 5). Onvansertib dose will be escalated in successive cohorts until the recommended phase 2 dose is achieved.
  Interventions: Drug: Onvansertib; Drug: Decitabine
- Phase 2: Onvansertib + decitabine (Experimental): Onvansertib recommended phase 2 dose, orally Day 1 through Day 5 every 28 days (1 cycle) and decitabine, administered consistently as 20 mg/m^2 intravenously over 1 hour on Day 1 through Day 5 every 28 days (1 cycle), with treatment modifications or delays based on return of hematopoietic function to baseline or Grade ≤1 toxicity for optimal subject management.
  Interventions: Drug: Onvansertib; Drug: Decitabine

INTERVENTIONS:
Drug: Onvansertib — Onvansertib orally
Drug: Cytarabine — subcutaneously
  Arms: Phase 1b: Onvansertib + low-dose cytarabine
Drug: Decitabine — intravenously
  Arms: Phase 1b: Onvansertib + decitabine; Phase 2: Onvansertib + decitabine

SUMMARY:
The purpose of the phase 1b/2 study is to determine whether Onvansertib given orally daily for 5 consecutive days every 28 days is safe and tolerable in adult patients who have relapsed/refractory Acute Myeloid Leukemia (AML), or are ineligible for intensive induction therapy, and to determine the maximum tolerated dose and recommended phase 2 dose of Onvansertib in combination with decitabine or Onvansertib in combination with low-dose cytarabine. In the phase 2 portion of the study, Onvansertib in combination with decitabine will be studied to provide further data on the safety profile of the combination and to preliminarily assess the activity of the chosen combination in patients with untreated AML who are not candidates for aggressive induction therapy, or who have received one prior treatment for their AML.

ELIGIBILITY:
Inclusion Criteria:

1. Disease Status and Prior Therapy:

   1. Histologically confirmed AML with >20% blasts
   2. Phase 1b: Participants with AML who are refractory to or have relapsed after initial treatment for their disease, with no more than three prior lines of therapy. Participants who have received prior treatment with cytarabine or decitabine are not excluded.
   3. Phase 2:

   i. Participants with AML who are refractory to, or have relapsed after, initial treatment for their disease, with no more than one prior line of therapy, and are judged not to be candidates for re-induction therapy that includes hematopoietic cell transplantation. Participants who have received prior cytarabine or decitabine are not excluded.

   OR

   ii. Participants with newly diagnosed, untreated AML ineligible for, or who have refused, standard intensive induction therapy
2. Age ≥18 years
3. ECOG performance status ≤2
4. Participants must be willing and able to review, understand, and provide written consent before starting any study-specific procedures or therapy.
5. All men and women must agree to practice effective contraception during the entire study period and after discontinuing study drug, unless documentation of infertility exists

   1. Sexually active, fertile women must use two effective forms of contraception (abstinence, intrauterine device, oral contraceptive, or double barrier device) from the time of informed consent and until at least 6 months after discontinuing study drug
   2. Sexually active men and their sexual partners must use effective contraceptive methods from the time of participant informed consent and until at least 3 months after discontinuing study drug

Exclusion Criteria:

1. Treatment-related AML or acute promyelocytic leukemia (APL)
2. Active malignancies within 12 months with the exception of those with a negligible risk of metastasis or death
3. Clinical evidence of active central nervous system leukemia at the time of screening
4. Alanine aminotransferase and/or aspartate aminotransferase ≥2.5 x upper limit of normal (ULN)
5. Total bilirubin > 2.0 mg/dL (or > 3.0 mg/dL in participants with documented Gilbert syndrome)
6. Serum creatinine ≥2.0 mg/dL
7. New York Heart Association Class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition, or hypertensive or metabolic condition
8. Myocardial infarction in the previous 12 weeks (from the start of treatment)
9. Resting left ventricular ejection fraction <50% at the time of screening
10. QT (Interval from the beginning of the QRS complex to the end of the T wave on an electrocardiogram) interval with Fridericia's correction [QTcF] >450 milliseconds. The QTcF should be calculated as the arithmetic mean of the QTcF on triplicate ECGs. In the case of potentially correctible causes of QT prolongation (e.g., medications, hypokalemia), the triplicate ECG may be repeated once during screening and that result may be used to determine eligibility.
11. Active and uncontrolled disease (other than AML) or infection as judged by the treating physician
12. Treatment with systemic therapy for the primary disease within 14 days (except for hydroxyurea or isolated doses of cytarabine or decitabine for white blood cell control)
13. Grade 2 or greater toxicities from prior therapy, except for Grade 2 toxicities that are not expected to resolve and that in the judgment of the Investigator do not pose a significant safety risk to subject participation.
14. Participants with any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the participant's ability to sign the informed consent form or his/her ability to cooperate and participate in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California Los Angeles, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - University of Kansas Cancer Center, Westwood, Kansas
  - Allina Health Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hagege A, Ambrosetti D, Boyer J, Bozec A, Doyen J, Chamorey E, He X, Bourget I, Rousset J, Saada E, Rastoin O, Parola J, Luciano F, Cao Y, Pages G, Dufies M. The Polo-like kinase 1 inhibitor onvansertib represents a relevant treatment for head and neck squamous cell carcinoma resistant to cisplatin and radiotherapy. Theranostics. 2021 Sep 21;11(19):9571-9586. doi: 10.7150/thno.61711. eCollection 2021. PMID 34646387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 participants were enrolled across 8 sites in the United States.
Groups:
- Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine: Participants were administered escalating doses of onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with cytarabine at a dose of 20mg/m^2 once daily on Day 1 up to Day 10 of each cycle, in order to determine the recommended phase 2 dose (RP2D) of onvansertib.
- Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine: Participants were administered escalating doses of onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with cytarabine at a dose of 20mg/m^2 once daily on Day 1 up to Day 10 of each cycle, in order to determine the RP2D of onvansertib.
- Phase 1b: Onvansertib 12 mg/m^2 + Decitabine; Phase 1b: Onvansertib 18 mg/m^2 + Decitabine; Phase 1b: Onvansertib 27 mg/m^2 + Decitabine; Phase 1b: Onvansertib 40 mg/m^2 + Decitabine; Phase 1b: Onvansertib 60 mg/m^2 + Decitabine; Phase 1b: Onvansertib 90 mg/m^2 + Decitabine: Participants were administered escalating doses of onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with decitabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle, in order to determine the RP2D of onvansertib.
- Phase 2: Onvansertib 60 mg/m^2 + Decitabine: Participants were administered onvansertib at the RP2D on Day 1 up to Day 5 of each cycle (where each cycle is 28 days), in combination with decitabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle.
Period: Overall Study
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine
Started | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6 | 32
Completed | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 4
Not Completed | 3 | 2 | 2 | 1 | 5 | 3 | 3 | 2 | 4 | 3 | 5 | 28
Not completed — Death | 2 | 2 | 2 | 1 | 4 | 2 | 2 | 2 | 3 | 3 | 4 | 24
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Safety/Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine: Participants were administered escalating doses of onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with cytarabine at a dose of 20mg/m^2 once daily on Day 1 up to Day 10 of each cycle, in order to determine the RP2D of onvansertib.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6 | 32 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 2 | 2 | 4 | 18
  >=65 years | 3 | 1 | 2 | 2 | 5 | 1 | 2 | 2 | 3 | 1 | 4 | 28 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 3 | 13 | 25
  Male | 3 | 2 | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 19 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5
  Not Hispanic or Latino | 3 | 1 | 3 | 3 | 4 | 4 | 3 | 1 | 4 | 1 | 6 | 30 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 6
  White | 2 | 2 | 3 | 3 | 4 | 4 | 3 | 1 | 4 | 2 | 5 | 29 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLT)
Description: Dose-limiting toxicities were defined as events related to onvansertib that were considered an adverse reaction or suspected adverse reaction during the first cycle of therapy and that fulfilled one of the following: Hematologic (persistent pancytopenia resistant to current standards of care that continues for ≥42 days and is not related to leukemic infiltration or another cause unrelated to study therapy) or Non-Hematologic (any Grade 3 abnormalities that persist >7 days without decreasing in severity despite standards of care, are clinically significant, or that are Grade 4 and symptomatic).
Time Frame: Up to Day 28 of Cycle 1
Population: The safety analysis set was comprised of all subjects who received at least one dose of onvansertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Statistical Analysis 1: Comparison: Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine vs Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine vs Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine vs Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine vs Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine vs Phase 1b: Onvansertib 12 mg/m^2 + Decitabine vs Phase 1b: Onvansertib 18 mg/m^2 + Decitabine vs Phase 1b: Onvansertib 27 mg/m^2 + Decitabine vs Phase 1b: Onvansertib 40 mg/m^2 + Decitabine vs Phase 1b: Onvansertib 60 mg/m^2 + Decitabine vs Phase 1b: Onvansertib 90 mg/m^2 + Decitabine; Test type: Other; Maximum Tolerated Dose = 60

2. Primary Outcome: Number of Participants With Change From Baseline in Eastern Co-operative Oncology Group (ECOG) Performance Status
Description: ECOG performance status was determined using 6-point scale from 0-5, with 0 meaning a participant was fully active/able to carry on all pre-disease activities without restriction and 5 meaning the participant was deceased.
Time Frame: Baseline and end of study (approximately up to up to 27 months)
Population: Per SAP It was pre-planned to report this data by treatment type instead of by dose.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Onvansertib + Low-dose Cytarabine: Participants were administered escalating doses of Onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with cytarabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle, in order to determine the recommended phase 2 dose (RP2D) of Onvansertib.
- Phase 1b: Onvansertib + Decitabine: Participants were administered escalating doses of Onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with decitabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle, in order to determine the recommended phase 2 dose (RP2D) of Onvansertib.
- Phase 2: Onvansertib + Decitabine: Participants were administered Onvansertib at the recommended phase 2 dose (RP2D) on Day 1 up to Day 5 of each cycle (where each cycle is 28 days), in combination with decitabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle.
Arm/Group | Phase 1b: Onvansertib + Low-dose Cytarabine | Phase 1b: Onvansertib + Decitabine | Phase 2: Onvansertib + Decitabine
Number analyzed (Participants) | 17 | 23 | 32
Participants | 11 | 14 | 22

3. Primary Outcome: Phase 2: Number of Participants Who Achieved a Complete Response (CR)
Description: Complete Response also includes Complete Response with Incomplete Blood Count Recovery (CRi). Complete response is defined by the following criteria:
  Morphologic leukemia-free state plus:
  * Subject is independent of transfusions
  * Absolute neutrophil count of >1000/mm3
  * Platelets of ≥100,000/mm3
  Complete response with incomplete blood count recovery meets all criteria for CR except for either neutropenia (ANC <1000/mm3) or thrombocytopenia (<100,000/mm3) but must include transfusion independence.
Time Frame: Up to 27 months
Population: Only participants in Phase 2 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Onvansertib + Decitabine
Number analyzed (Participants) | 32
Participants | 3

4. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Any clinically significant change in electrocardiogram (ECG), physical examination findings, body weight, vital signs, and laboratory parameters were recorded as Adverse Events.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 27 months)
Population: The safety analysis set was comprised of all subjects who received at least one dose of onvansertib.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Onvansertib 12 mg/m^2 + Decitabine; Phase 1b: Onvansertib 18 mg/m^2 + Decitabine; Phase 1b: Onvansertib 27 mg/m^2 + Decitabine; Phase 1b: Onvansertib 40 mg/m^2 + Decitabine; Phase 1b: Onvansertib 60 mg/m^2 + Decitabine; Phase 1b: Onvansertib 90 mg/m^2 + Decitabine: Participants were administered escalating doses of onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with decitabine at a dose of 20mg/m^2 once daily on Day 1 up to day 5 of each cycle, in order to determine the RP2D of Onvansertib.
- Phase 2: Onvansertib 60 mg/m^2 + Decitabine: Participants were administered onvansertib on Day 1 through Day 5 every 21 to 28 days, in combination with decitabine, administered consistently as 20 mg/m^2 over 1 hour on Day 1 through Day 5 every 28 days.
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6 | 32
Participants
  Any Adverse Events | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6 | 32
  Any Serious Adverse Events | 2 | 3 | 1 | 2 | 3 | 2 | 3 | 3 | 4 | 2 | 5 | 27
  Any Treatment-Related Serious Adverse Events | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 5

5. Secondary Outcome: Phase 2: Number of Participants Who Achieved a Morphologic Leukemia-free (MLF) State
Description: Defined as bone marrow (BM) <5% blasts in an aspirate with spicules and no blasts with Auer rods or persistence of extramedullary disease.
Time Frame: Up to 27 months
Population: Only participants in Phase 2 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Onvansertib + Decitabine
Number analyzed (Participants) | 32
Participants | 1

6. Secondary Outcome: Phase 2: Number of Participants With Partial Response (PR)
Description: PR criteria includes all of the hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate and a normalization of blood counts.
Time Frame: Up to 27 months
Population: Only participants included in Phase 2 were used in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Onvansertib + Decitabine
Number analyzed (Participants) | 32
Participants | 0

7. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: Duration of Response (DOR) is the time (in months) from the first response of CR, CRi or PR until recurrence of or progression of disease (or death). MLF State is also included as a response when calculating DOR. Responding subjects without death or progression will be censored at the date of their last evaluable disease assessment.
Time Frame: Up to 27 months
Population: Only participants in Phase 2 were included in this analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Onvansertib + Decitabine
Number analyzed (Participants) | 3
months | 5.2 [0.0 to 9.1]

8. Secondary Outcome: Phase 2: Event-free Survival (EFS)
Description: EFS is defined as the time from enrollment until disease progression or death from any cause and reported as the proportion of participants event free at 12 months.
Time Frame: 12 Months
Population: Only participants in Phase 2 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Phase 2: Onvansertib + Decitabine
Number analyzed (Participants) | 32
Proportion of Participants | 0.1 [0.0 to 0.2]

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the time from enrollment until death from any cause and reported as the proportion of participants alive at 12 months.
Time Frame: 12 Months
Population: Only participants included in Phase 2 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Phase 2: Onvansertib + Decitabine
Number analyzed (Participants) | 32
Proportion of Participants | 0.2 [0.1 to 0.4]

10. Secondary Outcome: Pharmacokinetic Parameter: Maximum Observed Plasma Concentration (Cmax) for Onvansertib
Time Frame: Cycle 1: Days 1 and 5
Population: The PK analysis set consisted of all subjects in the safety analysis set who received onvansertib and had adequate plasma onvansertib concentration data as determined by the PK scientist.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6 | 31
ng/mL
  Cycle 1 Day 1 | 92.57 (5.66) | 69.56 (28.73) | 251.16 (85.37) | 256.11 (24.96) | 626.18 (61.37) | 80.15 (21.33) | 129.18 (93.78) | 309.86 (72.47) | 410.42 (26.38) | 724.76 (57.33) | 737.21 (43.06) | 515.63 (43.47)
  Cycle 1 Day 5 | 139.22 (55.12) | 103.27 (43.01) | 298.63 (66.58) | 339.52 (31.25) | 857.29 (38.54) | 146.10 (56.75) | 197.67 (85.14) | 398.38 (32.95) | 496.24 (52.72) | 955.59 (54.78) | 1137.16 (61.56) | 861.86 (46.68)

11. Secondary Outcome: Pharmacokinetic Parameter: Time to Reach the Maximum Observed Plasma Concentration (Tmax) for Onvansertib
Time Frame: Cycle 1: Days 1 and 5
Population: as for outcome 10
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6 | 29
Hours
  Cycle 1 Day 1 | 1.961 (81.664) | 2.548 (96.282) | 2.301 (84.217) | 1.384 (103.829) | 2.071 (39.570) | 3.102 (31.792) | 2.365 (78.396) | 1.288 (41.249) | 1.373 (49.676) | 2.893 (135.893) | 2.435 (53.682) | 2.725 (69.661)
  Cycle 1 Day 5 | 1.844 (62.646) | 2.892 (37.244) | 2.267 (82.486) | 1.474 (67.999) | 2.148 (55.159) | 2.438 (24.524) | 1.583 (96.305) | 3.145 (33.877) | 3.161 (41.350) | 3.161 (41.350) | 3.189 (29.775) | 2.665 (51.333)

12. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Curve Over the First 24 Hours AUC(0-24) for Onvansertib
Time Frame: Cycle 1: Days 1 and 5
Population: as for outcome 10
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 6 | 32
h*ng/mL
  Cycle 1 Day 1 | 1197.93 (23.42) | 772.68 (26.21) | 2534.22 (31.05) | 2761.11 (36.97) | 5386.69 (59.16) | 1099.43 (29.81) | 2789.81 (25.30) | 3257.57 (53.53) | 4084.18 (27.94) | 9599.19 (25.01) | 9087.77 (57.43) | 6280.28 (46.85)
  Cycle 1 Day 5 | 1868.69 (70.99) | 3626.44 (5.33) | 5343.01 (2.11) | 7415.04 (64.35) | 19470.17 (17.10) | 1868.69 (70.99) | 3626.44 (5.33) | 5343.01 (2.11) | 7415.04 (64.35) | 19470.17 (17.10) | 12981.17 (56.18) | 11767.29 (39.78)

13. Secondary Outcome: Pharmacokinetic Parameter: Plasma Terminal Elimination Half-life (t1/2) for Onvansertib
Time Frame: Cycle 1: Days 1 and 5
Population: as for outcome 10
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 5 | 2 | 2 | 3 | 4 | 2 | 3 | 22
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 1 | 2 | 3 | 5 | 2 | 2 | 3 | 4 | 2 | 3 | 22
  Cycle 1 Day 1 | 11.294 (11.098) | 7.993 (NA) — Not calculable due to only 1 participant being analyzed. | 12.197 (71.258) | 11.747 (63.901) | 7.309 (99.539) | 16.960 (54.430) | 13.795 (28.866) | 9.394 (20.598) | 11.389 (39.530) | 12.917 (41.715) | 12.633 (50.655) | 11.904 (29.602)
  Cycle 1 Day 5: number analyzed (Participants) | 2 | 2 | 2 | 3 | 5 | 2 | 2 | 3 | 4 | 1 | 3 | 22
  Cycle 1 Day 5 | 16.413 (28.186) | 12.561 (38.983) | 12.246 (38.286) | 7.321 (8.094) | 14.484 (32.002) | 13.282 (39.361) | 9.082 (25.356) | 10.713 (23.782) | 16.337 (27.365) | 44.018 (NA) — Not calculable due to only 1 participant being analyzed. | 12.378 (10.948) | 14.060 (28.874)

ADVERSE EVENTS:
Time Frame: 27 months
Description: Participants included in the Safety Analysis Set were included in this analysis.
Groups:
- Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine; Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine: Participants were administered escalating doses of onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with cytarabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle, in order to determine the recommended phase 2 dose (RP2D) of onvansertib.
- Phase 1b: Onvansertib 12 mg/m^2 + Decitabine; Phase 1b: Onvansertib 18 mg/m^2 + Decitabine; Phase 1b: Onvansertib 27 mg/m^2 + Decitabine; Phase 1b: Onvansertib 40 mg/m^2 + Decitabine; Phase 1b: Onvansertib 60 mg/m^2 + Decitabine; Phase 1b: Onvansertib 90 mg/m^2 + Decitabine: Participants were administered escalating doses of onvansertib starting at 12mg/m^2 on Day 1 up to Day 5 of each cycle (where each cycle is 28 days) in combination with decitabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle, in order to determine the recommended phase 2 dose (RP2D) of onvansertib.
- Phase 2: Onvansertib 60 mg/m^2 + Decitabine: Participants were administered onvansertib at the recommended phase 2 dose (RP2D) on Day 1 up to Day 5 of each cycle (where each cycle is 28 days), in combination with decitabine at a dose of 20mg/m^2 once daily on Day 1 up to day 10 of each cycle.
Arm/Group | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine | Phase 2: Onvansertib 60 mg/m^2 + Decitabine
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 1/3 | 4/5 | 2/4 | 2/3 | 2/3 | 3/4 | 3/3 | 4/6 | 24/32
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 1/3 | 2/3 | 3/5 | 2/4 | 3/3 | 3/3 | 4/4 | 2/3 | 5/6 | 27/32
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 5/5 | 4/4 | 3/3 | 3/3 | 4/4 | 3/3 | 6/6 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine (N=5) | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine (N=4) | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine (N=3) | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine (N=3) | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine (N=4) | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine (N=3) | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine (N=6) | Phase 2: Onvansertib 60 mg/m^2 + Decitabine (N=32)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (4) | 1 (1) | 5 (10) | 8 (8)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Leukaemic infiltration pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Granulicatella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serratia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Onvansertib 12 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 18 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 27 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 40 mg/m^2 + Low-dose Cytarabine (N=3) | Phase 1b: Onvansertib 60 mg/m^2 + Low-dose Cytarabine (N=5) | Phase 1b: Onvansertib 12 mg/m^2 + Decitabine (N=4) | Phase 1b: Onvansertib 18 mg/m^2 + Decitabine (N=3) | Phase 1b: Onvansertib 27 mg/m^2 + Decitabine (N=3) | Phase 1b: Onvansertib 40 mg/m^2 + Decitabine (N=4) | Phase 1b: Onvansertib 60 mg/m^2 + Decitabine (N=3) | Phase 1b: Onvansertib 90 mg/m^2 + Decitabine (N=6) | Phase 2: Onvansertib 60 mg/m^2 + Decitabine (N=32)
Fatigue (General disorders) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 8 (8)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (6)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 9 (10)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 7 (9)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 2 (3) | 3 (5) | 9 (10)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (5)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 7 (9)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 | 2 (4) | 3 (3)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (4) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 2 (3) | 2 (2) | 4 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (3) | 2 (2) | 3 (7) | 1 (1) | 5 (10) | 12 (14)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 6 (9)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 3 (3)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (3)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Leukaemic infiltration pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Purpora (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 10 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03303339/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT03303339/SAP_001.pdf